CLINICAL TRIAL: NCT07373340
Title: A Pilot Randomized Clinical Study Comparing Patient-Reported Outcomes and Complications for Mandibular Implant Overdentures Retained by Different Splinted Attachment Systems
Acronym: M15011122
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Wageh Abozaed Elsaed Mansour, Principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15011122; M15011122 (Registry Identifier: Mansoyra university)
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Edentulism
Keywords: implant; overdenture; bar
MeSH Terms: interventions — Denture, Overlay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (bar locator): Patients were given overdentures with bar locator attachments, (Other)
  Interventions: Other: overdentures with bar locator attachments
- Group2: Patients were given overdentures with bar ball attachments (Other)
  Interventions: Other: overdentures with bar ball attachments

INTERVENTIONS:
Other: overdentures with bar locator attachments — Patients were given overdentures with bar locator attachments
  Arms: Group I (bar locator): Patients were given overdentures with bar locator attachments,
Other: overdentures with bar ball attachments — Patients were given overdentures with bar ball attachments
  Arms: Group2: Patients were given overdentures with bar ball attachments

SUMMARY:
This exploratory pilot randomized clinical study enrolled ten completely edentulous participants who experienced retention and stability problems with conventional mandibular complete dentures. Participants were randomly allocated to receive mandibular implant-supported overdentures retained by either a bar-locator attachment system (n = 5) or a bar-ball attachment system (n = 5). Denture satisfaction was assessed using the McGill Denture Satisfaction Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria incomplete mandibular edentulism for at least one year, adequate bone volume in the interforaminal region to permit implant placement, a documented history of insufficient retention and/or stability with a conventional mandibular complete denture.

Exclusion Criteria:

comprised uncontrolled systemic diseases, previous radiotherapy to the head and neck region, severe parafunctional habits, and any medical or local contraindications to implant surgery.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
patient-reported outcomes | Patient satisfaction (primary outcome) at T0 and after 6 months of overdenture insertion
  Patient satisfaction (primary outcome) between bar locator and bar ball using a McGill-based study at T0 and after 6 months of overdenture insertion
complications | prosthetic complication was evaluated From enrollment to the end of treatment at 3 years
  prosthetic complication between bar locator and bar ball

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Wageh, Al Mansurah, Egypt